CLINICAL TRIAL: NCT04684953
Title: Implantation of Thyroid Gland After Total Thyroidectomy in Quadriceps Femoris Muscle
Brief Title: Thyroid Autotransplantation in Quadriceps Femoris Muscle
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Hassan Aly, Resident surgeon, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: thyroid autotransplantation
Record Dates: First submitted 2020-12-22; First posted 2020-12-28 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Thyroid
MeSH Terms: conditions — Thyroid Diseases | interventions — Hormones

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thyroid autotransplantation (Active Comparator): Implantation of 5-10 gm thyroid gland after mincing it in saline in quadriceps femoris muscle.
  Interventions: Procedure: Throid autotransplantation
- control group (Other): the patients in this group won't undergo thyroid autotransplantation. instead, hormonal replacement therapy shall be prescribed for them.
  Interventions: Drug: Hormone

INTERVENTIONS:
Procedure: Throid autotransplantation — Operative
  Arms: Thyroid autotransplantation
Drug: Hormone — thyroid hormone replacement therapy
  Arms: control group

SUMMARY:
providing an almost natural ectopic thyroid in patients undergoing total thyroidectomy, remains a challenging subject that can benefits patients with a non-pharmacological substitute for their normal gland. this study seeks to prove that thyroid autotransplantation is possible and reliable.

DETAILED DESCRIPTION:
Total thyroidectomy, rather thyroidectomy, is currently widely accepted as the modality of choice for treatment of benign thyroid disorders that require surgical excision. The goal of post-thyroidectomy management is to reach a "safe physiological status" of thyroid hormonal profile. Although exogenous levothyroxine replacement has long been safely used as a replacement after total thyroidectomy, it is not considered optimal, as it is bounded by patient's compliance with the treatment and follow-up schedule, effect of mal-absorption, and the inability to compensate for daily physiological alterations.

The concept of endocrinal tissue auto-transplantation has been largely investigated in the case of parathyroid gland, and to a lesser extent for pancreatic islets. Although both the experimental studies of thyroid autotransplantation and the early case reports of lingual thyroid autotransplantations have shown encouraging results, a very limited number of clinical studies investigated thyroid autotransplantation in adult patients with benign thyroid disorders. Moreover, the discrepancy in the patients' characteristics and thyroid autotransplantation technique in these studies hinders the standardization of thyroid autotransplantation for clinical practice. Hypothetically, thyroid autotransplantation offers and attractive alternative for subtotal thyroidectomy, as it enables the preservation of native responsive thyroid tissue in an accessible location, and, thus, evades the risk of possible regrowth in the neck region. The present preliminary clinical study is conducted to investigate the feasibility and outcome of thyroid autotransplantation after total thyroidectomy for patients with benign thyroid disorders (other than thyroiditis).

ELIGIBILITY:
Inclusion Criteria:

* adult male or female with simple nodular goitre.
* patients who are fit for surgery.

Exclusion Criteria:

* children (male or female)
* patients with malignant or recurrent goitre
* patients who are unfit for surgery

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
normal level of thyroid hormone, and thyroid stimulating hormone | One year

CONTACTS AND LOCATIONS:
Overall Officials: Abdullah Badawy, professor, Study Director — general surgery professor; Ashraf Helmy, professor, Study Chair — general surgery professor; Mohamed M Saad Elshafey, professor, Study Chair — general surgery professor; Mohamed A Hassan, resident, Principal Investigator — resident physician at general surgery

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agarwal G, Aggarwal V. Is total thyroidectomy the surgical procedure of choice for benign multinodular goiter? An evidence-based review. World J Surg. 2008 Jul;32(7):1313-24. doi: 10.1007/s00268-008-9579-8. PMID 18449595
- [Background] Tominaga Y, Uchida K, Haba T, Katayama A, Sato T, Hibi Y, Numano M, Tanaka Y, Inagaki H, Watanabe I, Hachisuka T, Takagi H. More than 1,000 cases of total parathyroidectomy with forearm autograft for renal hyperparathyroidism. Am J Kidney Dis. 2001 Oct;38(4 Suppl 1):S168-71. doi: 10.1053/ajkd.2001.27432. PMID 11576947
- [Background] Wu Q, Zhang M, Qin Y, Jiang R, Chen H, Xu X, Yang T, Jiang K, Miao Y. Systematic review and meta-analysis of islet autotransplantation after total pancreatectomy in chronic pancreatitis patients. Endocr J. 2015;62(3):227-34. doi: 10.1507/endocrj.EJ14-0510. Epub 2015 Jan 7. PMID 25735805
- [Background] Papaziogas B, Antoniadis A, Lazaridis Ch, Makris J, Kotakidou R, Paraskevas G, Papaziogas T. Functional capacity of the thyroid autograft: an experimental study. J Surg Res. 2002 Apr;103(2):223-7. doi: 10.1006/jsre.2001.6348. PMID 11922738
- [Background] Shimizu K, Kumita S, Kitamura Y, Nagahama M, Kitagawa W, Akasu H, Oshina T, Kumasaki T, Tanaka S. Trial of autotransplantation of cryopreserved thyroid tissue for postoperative hypothyroidism in patients with Graves' disease. J Am Coll Surg. 2002 Jan;194(1):14-22. doi: 10.1016/s1072-7515(01)01115-2. PMID 11800336
- [Background] Al-Samarrai AY, Crankson SJ, Al-Jobori A. Autotransplantation of lingual thyroid into the neck. Br J Surg. 1988 Mar;75(3):287. doi: 10.1002/bjs.1800750333. No abstract available. PMID 3349341
- [Background] Swan H, Jenkins D, Schemmel J. Thyroid autograft. A 12-year follow-up. Arch Surg. 1967 Jun;94(6):817-20. doi: 10.1001/archsurg.1967.01330120071014. No abstract available. PMID 4226078
- [Background] Mohsen AA, Nada AA, Ibrahim MY, Ghaleb AH, Abou-Gabal MA, Mohsen AA, Wassef AT. Technique and outcome of autotransplanting thyroid tissue after total thyroidectomy for simple multinodular goiters. Asian J Surg. 2017 Jan;40(1):17-22. doi: 10.1016/j.asjsur.2015.05.007. Epub 2015 Aug 31. PMID 26337375
- [Background] Okamoto T, Fujimoto Y, Obara T, Ito Y, Kodama T, Kusakabe K. Trial of thyroid autotransplantation in patients with Graves' disease whose remnant thyroid has unintentionally been made too small at subtotal thyroidectomy. Endocrinol Jpn. 1990 Feb;37(1):95-101. doi: 10.1507/endocrj1954.37.95. PMID 2384054
- [Background] Roy PG, Saund MS, Thusoo TK, Roy D, Sankar R. Fate of human thyroid tissue autotransplants. Surg Today. 2003;33(8):571-6. doi: 10.1007/s00595-003-2557-8. PMID 12884093
- [Background] Sheverdin IuP. [The results of a 15-year observation of patients with an autotransplant of thyroid gland fragments performed to prevent postoperative hypothyroidism]. Vestn Khir Im I I Grek. 1992 Feb;148(2):152-6. Russian. PMID 8594711
- [Background] Ozdemir D, Cuhaci FN, Ozdemir E, Aydin C, Ersoy R, Turkolmez S, Cakir B. The role of postoperative Tc-99m pertechnetate scintigraphy in estimation of remnant mass and prediction of successful ablation in patients with differentiated thyroid cancer. Nucl Med Commun. 2016 Jun;37(6):640-5. doi: 10.1097/MNM.0000000000000492. PMID 26895488
- [Background] Uzzan B, Campos J, Cucherat M, Nony P, Boissel JP, Perret GY. Effects on bone mass of long term treatment with thyroid hormones: a meta-analysis. J Clin Endocrinol Metab. 1996 Dec;81(12):4278-89. doi: 10.1210/jcem.81.12.8954028.
- [Result] Katna R, Kalyani N, Deshpande A; Mumbai Oncology Group - Head and Neck. Free thyroid transfer to anterolateral thigh for prevention of radiation induced hypothyroidism: An initial experience. Am J Otolaryngol. 2019 Mar-Apr;40(2):160-163. doi: 10.1016/j.amjoto.2018.12.013. Epub 2018 Dec 21. PMID 30594401